CLINICAL TRIAL: NCT05490745
Title: A Psychological Intervention for Children's Mental Health Problems or Disorders Based on Parental Reflective Functioning to Enhance Positive Parenting During Adverse Situations
Brief Title: Psychological Intervention for Child Mental Health Based on Parental Reflective Functioning to Enhance Positive Parenting
Acronym: SK4Parenting+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other); Psychology Research Center (CIPsi) (Unknown); Psychology Association of the University of Minho (aPsi-UMinho) (Unknown); ProChild CoLAB - The Collaborative Laboratory against child poverty and social exclusion (Unknown)
Responsible Party: Principal Investigator, Bárbara Figueiredo, Associate Professor with Aggregation, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEICSH 106/2020; CIPSI-VC-2020-01 (Other Grant/Funding Number: Foundation for Science and Technology (FCT))
Record Dates: First submitted 2022-07-28; First posted 2022-08-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Externalizing Problems; Internalizing Problems
Keywords: Positive Parenting; Pre-school Children; Parents; Adversity; Psychological Problems; Parental Reflective Functioning; Psychological Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Waiting Lists; Nocebo Effect

STUDY DESIGN:
Intervention Model Description: The interventional model is a simple two-arm RCT study (intervention vs. waiting-list), with 3 to 4 assessment waves (Time 0, Time 0+, Time 1, Time 2).
  If the child is included in the study, they will be subject to a randomization process, being allocated, considering a sequence of random numbers generated by computer in a 1:1 ratio. In the randomization, half of the children are allocated to the IIG and the other half to the DIG.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Intervention Group (IIG) (Experimental): Participants receive initially one session for psychological assessment. At the end of the session, the second session is scheduled for the following week, where feedback about the assessment will be provided. If in the second session participants agree to proceed with the psychological intervention, then the remaining 4-6 sessions of Skills4Parenting+ are conducted.
  Interventions: Behavioral: Skills4Parenting+
- Delayed Intervention Group (DIG) (Other): Waiting-list Comparator (nocebo): Participants initially receive one session for psychological assessment. At the end of the session, participants are informed that they will be contacted to schedule the second session, where feedback about the assessment will be provided. Participants are contacted during the same week, to schedule the second session 8 weeks after the first session. If in the second session participants agree to proceed with the psychological intervention, then the remaining 4-6 sessions of Skills4Parenting+ are conducted.
  Interventions: Other: Waiting-list (nocebo)

INTERVENTIONS:
Behavioral: Skills4Parenting+ — Skills4Parenting+ has 6-8 weekly individual online sessions (50 min) + 8-week follow-up. First, an assessment session of parents' positive parenting skills (PPS), based on mother/father-child interaction observation. The following sessions aim to (1) promote parental reflective functioning, enhancing parents' understanding of the child´s problems, and (2) activate PPS to solve the child's problems. Written registers of problematic situations - in which the problems of the child occur, are analyzed (i.e., child's and parents' behaviors, thoughts, and feelings) (intersession activity) - are reflected upon, to understand and solve through PPS. PPS implementations are analyzed to understand the changes in the child and parent. Future situations and activation of appropriate PPS are anticipated, to solve potential upcoming problems of the child's, related to adversity. When the therapeutic goals have not been fully achieved, two additional sessions (total of 8 instead of 6), are added.
  Arms: Immediate Intervention Group (IIG)
Other: Waiting-list (nocebo) — Participants wait to receive the psychological intervention (Skills4Parenting+) for eight weeks, after the assessment session.
  Arms: Delayed Intervention Group (DIG)

SUMMARY:
In this study we aim to verify the effectiveness of a psychological intervention for preschool children, 3 to 6 years of age, with psychological problems or disorders, arising from adversity, Skills4Parenting+.

Skills4Parenting+, with 6 to 8 weekly sessions, aims to treat the child's psychological problems or disorders, based on parental reflective functioning, to activate and develop parents' positive parenting skills, in response to situations of adversity.

To assess the effectiveness, we plan to conduct an a simple two-arm RCT study, where children are randomly allocated to an immediate intervention group (IIG) or a delayed intervention group (DIG).

The IIG will be assessed at 3 time-points: Time 0 (pre-test: before the 1st session); Time 1 (post-test: after the last session) and Time 2 (follow-up: 8 weeks after the last session). The DIG will be assessed at 4 time-points: Time 0 (pre-test 1: before the 1st session); Time 0+ (pre-test 2: 8 weeks after the 1st session); Time 1 (post-test: after the last session) and Time 2 (follow up: 8 weeks after the last session). A time period of 8 weeks will be maintained between each time point.

In this study, we expect the (1) psychological intervention to significantly diminish the child's psychological problems or disorders (from pretest to posttest); (2) parental reflective functioning will mediate the effect of the psychological intervention on child's psychological problems or disorders; (3) the children from IIG will demonstrate a significant improvement in their mental health, in comparison to the children from the DIG; and (4) for the effects of the psychological intervention (i.e., improvement in the child's mental health) to be maintained in the medium-term (from posttest to follow-up).

DETAILED DESCRIPTION:
1. Introduction Due to the negative effects of adversity on child mental health and development [1], this study proposes a validation of a psychological intervention, Skills4Parenting+, which aims to respond to the mental health needs of preschool children (3 to 6 years of age), in a preventive and remedial manner. This intervention is based on strong empirical evidence, such as Positive parenting from zero to three, the "Online Parenting Pro-Tips (OPPT)" [2], and parental reflective functioning [3].
2. Aims The aim of this project is to implement and study the effectiveness of a psychological intervention, Skills4Parenting+, for children with psychological problems or disorder and their families, associated with situations of adversity.
3. Methodology 3.1. Participants The target population of this project are children, aged between 3 and 6 years, including those attending pre-school of the public school system of the Municipality of Guimarães, and from aPsi - Psychology Association of the University of Minho, and their parents, who hold parental responsibilities. If validated, the procedures of Skills4Parenting+ can be replicated in other community contexts.

Recruitment of participants is done through the websites: + Citizenship (https://maiscidadania.cim-ave.pt/), CIPsi (https://www.psi.uminho.pt/pt/CIPsi), ProChild CoLAB (http: / /prochildcolab.pt), APsi-UMinho (https://apsi.uminho.pt) and Guimarães City Hall (https://www.cm-guimaraes.pt), as well as through the social networks of these institutions. In addition, posters, in various locations in the Municipality of Guimarães, roll-ups in formal events, postcards, delivered to children and families, and information about the project will be disseminated in local newspapers and radio in the Municipality of Guimarães.

Participants of (1) the screening procedure who access the + Citizenship platform (https://maiscidadania.cim-ave.pt/) or (2) of aPsi are all those who are self-referred to the private psychological services of aPsi, who hold parental responsibilities of at least one child under the conditions mentioned above, consent to participate in the study after being informed of the goals and procedures, who answer the screening questionnaires and who meet eligibility criteria.

3.2. Assessment Procedures The child's and their family's psychological assessment aim to: (1) validate the conditions necessary to implement a psychological intervention and (2) guide the child's psychological intervention.

If the report from the child's legal guardian indicates, during the screening, signs of psychological problems or disorder in the child, the child's legal guardian is invited to complete the psychological assessment through questionnaires.

The psychological assessment is carried out mostly online and lasts approximately 40 minutes. The questionnaires are answered (1) on the ProChild platform integrated with the + Citizenship platform and the Child Behavior Checklist (CBCL) is sent and returned by mail or (2) delivered in person or via mail, in paper, through aPsi's services.

After the child's legal guardian filled out the respective questionnaires, the screening and assessment data are analyzed and synthesized in an evaluation report.

In order to start the selection of children and families, the child's legal guardian is contacted by telephone to make an initial appointment. Posteriorly, if the child meets eligibility criteria, the materials necessary to carry out the evaluation at the first session and Informed Consent are delivered. In this consent, the child's legal guardian is asked to authorize a) their participation and the child's participation in the psychological intervention phase, b) filing in questionnaires for the orientation and monitoring of the psychological intervention, c) the realization of online sessions, if necessary, d) the videorecording of sessions and e) the data provided in the questionnaires. The child's legal guardian, who consent to subparagraphs a) and b), but not subparagraphs c), d), e), or f) may benefit from psychological intervention, if this is their will.

3.3. Intervention Procedures The first intervention session consists of a psychological assessment, which aims to, among others, validate the conditions necessary for the implementation of a psychological intervention. The session is scheduled and carried out with at least one of the child's legal guardians, after being informed about the goals and procedures of the psychological intervention and signing the Informed Consent. This assessment session lasts 45 to 60 minutes. After consent of the child's legal guardian is given, the session is videorecorded.

The structure of this session consists of a clinical interview, directed to the parents, considering the elements resulting from the evaluation report.

If the child meets any of the exclusion criteria, they are not followed up under this Program and are referred to an appropriate service. For children who are not participating in the study, an online session will be scheduled to return the results and justify the exclusion and/or referral. For children who are included in the intervention, a randomized controlled trial (RCT) will be carried out. According to it, the next session can be scheduled for the following week (IIG) or up to eight weeks after the first session (DIG). Participants who wait eight weeks are informed of the telephone line and e-mail, which they can use if necessary.

Psychological intervention is carried out by psychologists duly accredited by the Order of Portuguese Psychologists (OPP). It is carried out online or in person according to the updates of the General Directorate of Health (DGS) recommendations, regarding the evolution of the pandemic.

3.4. Randomization and Monitoring This project considers a simple two-arm RCT with the aim of randomly allocating participants into two intervention groups (IIG, DIG) in order to assess the effectiveness of a psychological intervention in comparison to a waiting list. This waiting list also facilitates the management of resources for the intervention provided in this project.

Monitoring is also carried out (through responses to evaluation questionnaires) with the aims of (1) monitoring the situation of the child and the family awaiting psychological intervention, (2) monitoring the response of the child and the family to the intervention and (3) evaluate the effectiveness of the intervention programs provided.

In case the child is part of the psychological intervention, Skills4Parenting+, it will be subjected to a randomization process, being allocated to one of the two groups, considering a sequence of random numbers generated by the computer. In this randomization, half of the children will be allocated to the psychological intervention (IIG), while the other half to a waiting list (DIG; after eight weeks).

After the last session (6th or 8th session) of the psychological intervention, an assessment is performed in order to verify if the child shows significant improvements or if he/she remains with psychopathological symptoms. After the conclusion of the assessment, cases that present at least two of the following elements, are referred to a targeted therapy, specific to the child's problems: (1) SDQ higher than the cutoff point (≥16), (2) indication of one or more trauma items in SPAS, and (3) continued impact of the effects of the adverse situation.

After the end of the psychological intervention, a follow-up session will be held 8 weeks later.

3.5. Data analysis procedures At least 60 children and their families will be recruited within the scope of the proposed psychological intervention. With n ≥ 30 in each group (2 groups), the effectiveness study of psychological intervention has a power of + 95% to detect medium-to-high effects (sample size calculator for SMART designs; 4,5).

If missing data is verified during descriptive analysis, the data will be imputated (if percentage of missing data is low) or removed (if percentage of missing data is high).

The data will be analyzed using the statistical software SPSS version 27. The normality of the data will be verified through the Kolmogorov-Smirnov test.

Descriptive analyzes and tests of differences between groups will be carried out (T-test or non-parametric equivalent).

To assess the effectiveness of the intervention, an ANOVA and MANOVA of repeated measures will be conducted with the different outcome variables, with an intra-subject factor (evaluation moments: Time 0, Time 0+, Time 1, Time 2) and with factor between groups (IIG, DIH).

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 and 6 years old, inclusive
* Signaling in the screening (≥16 in the SDQ total scale)
* CBCL (i.e., ≥60 on the Internalizing and/or Externalizing Scale) OR Parents report a high pandemic impact
* Parental informed consent and commitment to the planned psychological intervention.
* Parent is the child's legal guardian

Exclusion Criteria:

* Already receiving psychological intervention
* Presence of psychological problems not related to an adverse situation or not likely to be monitored within the scope of the proposed intervention (for example, autism spectrum or intellectual development disorders or, domestic violence, neglect or abuse prior to the adverse situation);
* Do not speak or understand Portuguese

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change (Arm 1) "Strengths & Difficulties Questionnaire" (SDQ [6]; Portuguese version [7]) | 3 time-points: Time 0 (1-2 weeks before 1st session); Time 1 (1 week after last session); and Time 2 (8 weeks after last session).
  Questionnaire with 25 items that seek to assess emotional and behavioral problems, which can be answered by parents and teachers of children from 3 to 16 years old. In this study, only the version for parents is used. The items are scored on a 3-point scale (0 = "Not true", 1 = "It is a bit true" and "2 = It is very true"). It comprises five subscales: (1) emotional symptoms, (2) conduct problems, (3) hyperactivity, (4) peer problems and (5) prosocial behavior. The sum of the first four subscales (with the exception of the prosocial behavior scale) allows the calculation of the total of difficulties, which can vary between 0 and 40. In addition to the 25 items, 5 additional items are applied to assess the impact of the reported problems in the child's life. The cutoff point of the questionnaire is 16 or more points, on the total scale, indicating clinical level of the child's emotional and behavioral problems.
Change (Arm 1) "Child Behavior Checklist 1½-5 "(CBCL [8]; Portuguese version [9]) | 2 time-points: Time 0 (1-2 weeks before 1st session); and Time 2 (8 weeks after last session)
  Questionnaire composed of 113 items that assess internalizing (i.e., anxiety/depression, isolation, somatic complaints), externalizing (i.e., delinquent behavior, aggressive behavior), social, thinking and attention problems of the child. Each item is answered on a 3-point likert scale (0 = statement is not true to 2 = statement that is very true or often true).
Change (Arm 2) "Strengths & Difficulties Questionnaire" (SDQ [6]; Portuguese version [7]) | 4 time-points: Time 0 (1-2 weeks before 1st session); Time 0+ (8 weeks after Time 0); Time 1 (1 week after last session); and Time 2 (8 weeks after last session)
  Questionnaire with 25 items that seek to assess emotional and behavioral problems, which can be answered by parents and teachers of children from 3 to 16 years old. In this study, only the version for parents is used. The items are scored on a 3-point scale (0 = "Not true", 1 = "It is a bit true" and "2 = It is very true"). It comprises five subscales: (1) emotional symptoms, (2) conduct problems, (3) hyperactivity, (4) peer problems and (5) prosocial behavior. The sum of the first four subscales (with the exception of the prosocial behavior scale) allows the calculation of the total of difficulties, which can vary between 0 and 40. In addition to the 25 items, 5 additional items are applied to assess the impact of the reported problems in the child's life. The cutoff point of the questionnaire is 16 or more points, on the total scale, indicating clinical level of the child's emotional and behavioral problems.
Change (Arm 2) "Child Behavior Checklist 1½-5 "(CBCL [8]; Portuguese version [9]) | 2 time-points: Time 0 (1-2 weeks before 1st session); and Time 2 (8 weeks after last session)
  Questionnaire composed of 113 items that assess internalizing (i.e., anxiety/depression, isolation, somatic complaints), externalizing (i.e., delinquent behavior, aggressive behavior), social, thinking and attention problems of the child. Each item is answered on a 3-point likert scale (0 = statement is not true to 2 = statement that is very true or often true).

SECONDARY OUTCOMES:
Change (Arm 1) "COVID-19 Pandemic Impact Questionnaire" | 3 time-points: Time 0 (1-2 weeks before 1st session); Time 1 (1 week after last session); and Time 2 (8 weeks after last session).
  Questionnaire composed of 25 items that seek to assess the impact of covid-19 pandemic on the family, which can be answered by parents. Six items are scored on dichotomous scale, two items are scored on a 3-point scale, three items are scored on a 4-point scale, thirteen items are scored on a 5-point scale and one item is scored on a 6-point scale. It comprises five subscales: (1) health and covid-19 exposure, (2) family dynamics, (3) school, (4) social contact and (5) daily behaviors. The sum of the five subscales (with the exception of the prosocial behavior scale) allows the calculation of the total impact, which can vary between 0 and 86, with the impact being greater when the score is higher.
Change (Arm 1) "Spence Preschool Anxiety Scale" (SPAS [10]; Portuguese version [11]) | 3 time-points: Time 0 (1-2 weeks before 1st session); Time 1 (1 week after last session); and Time 2 (8 weeks after last session).
  Questionnaire applied to parents, consisting of 28 items that assess problems related to 5 types of anxiety disorders present in preschool age: Generalized anxiety, social anxiety, separation anxiety, fear of physical damage and obsessive-compulsive disorder. Six additional items assess the presence of post-traumatic stress disorder symptoms. Each item is answered using a 5-point likert scale (0 = never to 4 = always). The partial results and the overall result are calculated by the sum of the responses to the items.
Change (Arm 1) "Parental Practices Interview" (PPI [12]; Portuguese version [13]) | 3 time-points: Time 0 (1-2 weeks before 1st session); Time 1 (1 week after last session); and Time 2 (8 weeks after last session).
  Rigid and inconsistent Discipline Scale composed of 16 items, evaluated on a 7-point likert scale (1 = never to 7 = always). Higher scores are associated with more rigid and inconsistent parenting practices.
Change (Arm 1) "Parental Reflective Functioning Questionnaire" (PRFQ [14]; Portuguese version [15]) | 3 time-points: Time 0 (1-2 weeks before 1st session); Time 1 (1 week after last session); and Time 2 (8 weeks after last session).
  PRFQ is a 18-item self-report multidimensional questionnaire, scored on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). It was designed for parents of children aged 0 to 5 years to assess three key dimensions of PRF: an interest and curiosity in a child's mental states, the ability to recognize that a child's mental states may not be fully accessible, and difficulties with mentalization. The PRFQ comprises three subscales for assessing the abovementioned dimensions. The first subscale, Pre-Mentalizing Modes of Mental States (PM), Certainty about Mental States (CMS), Interest and Curiosity in Mental States (IC).
(Arm 1) "Brief Problem Monitor" (BPM [16]; Portuguese version in publication) | 1 time-point: Time 1 (1 week after last session).
  BPM is a reduced version of CBCL that is used to prevent/control the learning effect. This questionnaire consists of 19 items scored on a 3-point likert scale from 0 (not true) to 2 (very true) and aims to evaluate responses regarding clinical intervention with children, through regular monitoring of the therapeutic process.
"Skills4Parenting+ Satisfaction Questionnaire" | 1 time-point: Time 1 (1 week after last session; both arms)
  Questionnaire composed of 33 items that seek to assess the level of parental satisfaction with the program Skills4Parenting+. 26 items are scored on a 7-point likert scale and seven items are of open and optional response.
Change (Arm 2) "COVID-19 Pandemic Impact Questionnaire" | 4 time-points: Time 0 (1-2 weeks before 1st session); Time 0+ (8 weeks after Time 0); Time 1 (1 week after last session); and Time 2 (8 weeks after last session).
  Questionnaire composed of 25 items that seek to assess the impact of covid-19 pandemic on the family, which can be answered by parents. Six items are scored on dichotomous scale, two items are scored on a 3-point scale, three items are scored on a 4-point scale, thirteen items are scored on a 5-point scale and one item is scored on a 6-point scale. It comprises five subscales: (1) health and covid-19 exposure, (2) family dynamics, (3) school, (4) social contact and (5) daily behaviors. The sum of the five subscales (with the exception of the prosocial behavior scale) allows the calculation of the total impact, which can vary between 0 and 86, with the impact being greater when the score is higher.
Change (Arm 2) "Spence Preschool Anxiety Scale" (SPAS [10]; Portuguese version [11]) | 4 time-points: Time 0 (1-2 weeks before 1st session); Time 0+ (8 weeks after Time 0); Time 1 (1 week after last session); and Time 2 (8 weeks after last session).
  Questionnaire applied to parents, consisting of 28 items that assess problems related to 5 types of anxiety disorders present in preschool age: Generalized anxiety, social anxiety, separation anxiety, fear of physical damage and obsessive-compulsive disorder. Six additional items assess the presence of post-traumatic stress disorder symptoms. Each item is answered using a 5-point likert scale (0 = never to 4 = always). The partial results and the overall result are calculated by the sum of the responses to the items.
Change (Arm 2) "Parental Practices Interview" (PPI [12]; Portuguese version [13]) | 4 time-points: Time 0 (1-2 weeks before 1st session); Time 0+ (8 weeks after Time 0); Time 1 (1 week after last session); and Time 2 (8 weeks after last session).
  Rigid and inconsistent Discipline Scale composed of 16 items, evaluated on a 7-point likert scale (1 = never to 7 = always). Higher scores are associated with more rigid and inconsistent parenting practices.
Change (Arm 2) "Parental Reflective Functioning Questionnaire" (PRFQ [14]; Portuguese version [15]) | 4 time-points: Time 0 (1-2 weeks before 1st session); Time 0+ (8 weeks after Time 0); Time 1 (1 week after last session); and Time 2 (8 weeks after last session).
  PRFQ is a 18-item self-report multidimensional questionnaire, scored on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). It was designed for parents of children aged 0 to 5 years to assess three key dimensions of PRF: an interest and curiosity in a child's mental states, the ability to recognize that a child's mental states may not be fully accessible, and difficulties with mentalization. The PRFQ comprises three subscales for assessing the abovementioned dimensions. The first subscale, Pre-Mentalizing Modes of Mental States (PM), Certainty about Mental States (CMS), Interest and Curiosity in Mental States (IC).
Change (Arm 2) "Brief Problem Monitor" (BPM [16]; Portuguese version in publication) | 2 time-points: Time 0+ (8 weeks after Time 0); and Time 1 (1 week after last session)
  BPM is a reduced version of CBCL that is used to prevent/control the learning effect. This questionnaire consists of 19 items scored on a 3-point likert scale from 0 (not true) to 2 (very true) and aims to evaluate responses regarding clinical intervention with children, through regular monitoring of the therapeutic process.

OTHER OUTCOMES:
"Sociodemographic Questionnaire" | 1 time-point: Time 0 (1-2 weeks before 1st session; both arms).
  The Sociodemographic Questionnaire was used to collect sociodemographic information of the child and parents - such as gender, age, nationality, household members, socioeconomic level and schooling.
Change (Arm 1) "Warwick-Edinburgh Mental Well-Being Scale" (WEMWBS [17]; Portuguese version [18]) | 3 time-points: Time 0 (1-2 weeks before 1st session); Time 1 (1 week after last session); Time 2 (8 weeks after last session).
  Self-report scale composed of 14 items, scored on a 5-point likert scale (1= never to 5= always), to assess mental health and well-being. The minimum score is 14 points and the maximum score is 70 points, where the higher levels are associated with better mental well-being.
Change (Arm 2) "Warwick-Edinburgh Mental Well-Being Scale" (WEMWBS [17]; Portuguese version [18]) | 4 time-points: Time 0 (1-2 weeks before 1st session); Time 0+ (8 weeks after Time 0); Time 1 (1 week after last session); Time 2 (8 weeks after last session).
  Self-report scale composed of 14 items, scored on a 5-point likert scale (1= never to 5= always), to assess mental health and well-being. The minimum score is 14 points and the maximum score is 70 points, where the higher levels are associated with better mental well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minho, Braga, Braga District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ravens-Sieberer U, Kaman A, Erhart M, Devine J, Schlack R, Otto C. Impact of the COVID-19 pandemic on quality of life and mental health in children and adolescents in Germany. Eur Child Adolesc Psychiatry. 2022 Jun;31(6):879-889. doi: 10.1007/s00787-021-01726-5. Epub 2021 Jan 25. PMID 33492480
- [Background] [2] Riegler, L. J., Raj, S. P., Moscato, E. L., Narad, M. E., Kincaid, A., & Wade, S. L. (2020). Pilot trial of a telepsychotherapy parenting skills intervention for veteran families: Implications for managing parenting stress during COVID-19. Journal of Psychotherapy Integration, 30(2), 290. doi: 10.1037/int0000220
- [Background] Ensink K, Borelli JL, Roy J, Normandin L, Slade A, Fonagy P. Costs of Not Getting to Know You: Lower Levels of Parental Reflective Functioning Confer Risk for Maternal Insensitivity and Insecure Infant Attachment. Infancy. 2019 Mar;24(2):210-227. doi: 10.1111/infa.12263. Epub 2018 Oct 11. PMID 32677198
- [Background] [4] Crivello, A.I., Levy, J.A., & Murphy, S.A. 2007a. Evaluation of Sample Size Formulae for Developing Adaptive Treatment Strategies Using a SMART Design. Tech. rept. No. 07-81. University Park, PA: The Pennsylvania State University, The Methodology Center.
- [Background] [5] Crivello, A.I., Levy, J.A., & Murphy, S.A. 2007b. Statistical Methodology for a SMART Design in the Development of Adaptive Treatment Strategies. Tech. rept. No. 07-82. University Park, PA: The Pennsylvania State University, The Methodology Center.
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] [7] Fleitlich, B., Loureiro, M., Fonseca, A., & Gaspar, F. (2005). Questionário de capacidades e dificuldades (SDQ-Por)[Strengths and Difficulties Questionnaire, Portuguese version]. Retrived from http://www. sdqinfo. org.
- [Background] [8] Achenbach, T. M., & Rescorla, L. A. (2000). Manual for the ASEBA preschool forms and profiles (Vol. 30). Burlington, VT: University of Vermont, Research center for children, youth, & families.
- [Background] [9] Achenbach, T. M., Rescorla, L. A., Dias, P., Ramalho, V., Lima, V. S., Machado, B. C., & Gonçalves, M. (2014). Manual do sistema de avaliação empiricamente validado (ASEBA): Um sistema integrado de avaliação com múltiplos informadores. Manual do período pré-escolar e do período escolar. Braga: Psiquilibrios Edições
- [Background] Spence SH, Rapee R, McDonald C, Ingram M. The structure of anxiety symptoms among preschoolers. Behav Res Ther. 2001 Nov;39(11):1293-316. doi: 10.1016/s0005-7967(00)00098-x. PMID 11686265
- [Background] [11] Almeida, J. P., & Viana, V. (2013). Adaptação da escala de ansiedade pré-escolar, de s. Spence. Psicologia, Saúde & Doenças, 14(3), 470-483.
- [Background] Webster-Stratton C, Reid MJ, Hammond M. Preventing conduct problems, promoting social competence: a parent and teacher training partnership in head start. J Clin Child Psychol. 2001 Sep;30(3):283-302. doi: 10.1207/S15374424JCCP3003_2. PMID 11501247
- [Background] Sousa PM, Gaspar P, Fonseca H, Gaspar F. Association between treatment adherence and quality of life among overweight adolescents. Cad Saude Publica. 2017 Jan 23;33(1):e00171815. doi: 10.1590/0102-311X00171815. PMID 28125128
- [Background] Luyten P, Mayes LC, Nijssens L, Fonagy P. The parental reflective functioning questionnaire: Development and preliminary validation. PLoS One. 2017 May 4;12(5):e0176218. doi: 10.1371/journal.pone.0176218. eCollection 2017. PMID 28472162
- [Background] Moreira H, Fonseca A. Measuring Parental Reflective Functioning: Further Validation of the Parental Reflective Functioning Questionnaire in Portuguese Mothers of Infants and Young Children. Child Psychiatry Hum Dev. 2023 Aug;54(4):1042-1054. doi: 10.1007/s10578-021-01288-2. Epub 2022 Jan 22. PMID 35064394
- [Background] [16] Achenbach, T. M., McConaughy, S. H., Ivanova, M. Y., & Rescorla, L. A. (2011). Manual for the ASEBA brief problem monitor (BPM). Burlington, VT: ASEBA, 33
- [Background] [17] Stewart-Brown, S., & Janmohamed, K. (2008). Warwick-Edinburgh mental well-being scale. User guide. Version, 1(10.1037).
- [Background] [18] Alho, L. J. N. D. S. (2021). Pandemia COVID-19: bem-estar e saúde mental de profissionais da saúde e da educação (Doctoral dissertation).